CLINICAL TRIAL: NCT05024201
Title: The Effect Of Therapeutic Touch Applied to Hemodialysis Patient On The Level Of Loneliness And Hopelessness
Brief Title: The Effect Of Therapeutic Touch On Loneliness and Hopelessness
Acronym: nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zehra Bayram (Other)
Responsible Party: Sponsor-Investigator, Zehra Bayram, Nurse, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10364632
Record Dates: First submitted 2021-04-21; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: Loneliness; Hope
Keywords: Hemodialysis; Nursing; Loneliness; Hopelessness; Therapeutic Touch
MeSH Terms: interventions — Touch

STUDY DESIGN:
Intervention Model Description: In this study, two scales will be used to measure the loneliness and hopelessness levels of hemodialysis patients. Patients will fill in UCLA Loneliness Scale and BECK Hopelessness Scale.Therapeutic touch treatment method will provide nurses the holistic caregiver role for the feelings of loneliness and hopelessness experienced by the patients. When the literature is scanned, this study is unique because it has not been done before on hemodialysis patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group for effect of therapeutic touch (Experimental): Therapeutic touch was applied to the experimental group for three days every other day.
  Interventions: Behavioral: THERAPEUTİC TOUCH FOR HEMODİALYSİS PATİENTS
- control group for effect of therapeutic touch (No Intervention): No application was applied to the control group. Only pretest and posttest were done.

INTERVENTIONS:
Behavioral: THERAPEUTİC TOUCH FOR HEMODİALYSİS PATİENTS — Therapeutic touch was applied to hemodialysis patients for 3 days every other day.
  Arms: experimental group for effect of therapeutic touch

SUMMARY:
The effect of therapeutic touch applied to hemodialysis patients on the level of loneliness and hopelessness is being investigated. It encourages nurses to practice therapeutic touch.

DETAILED DESCRIPTION:
Chronic diseases are a challenging process that affects human life physiologically and psychologically. Chronic Renal Failure, which shows a significant increase in the world and in our country, also affects human life in every aspect. Hemodialysis treatment is used with a high rate in the treatment of patients diagnosed with End Stage Renal Failure.

Hemodialysis patients experience loneliness and hopelessness during their difficult and compulsory treatmet. Fear of being alone is an important problem affecting the patient's compliance with treatment. In addition, the other problem these patients experience is hopelessness. Hopelessness is an important factor that affects the patient's expectations for the future and the process of solving problems.

Therapeutic touch is a complementary and alternative treatment method. It is stated that this treatment method, which is successfully used by nurses, is good for loneliness and hopelessness. This method, which will be used on hemodialysis patients, is aimed to get away from the problems of loneliness and hopelessness.

In this study, two scales will be used to measure the loneliness and hopelessness levels of hemodialysis patients. Patients will fill in UCLA Loneliness Scale and BECK Hopelessness Scale.

Nurses should not ignore the problems of loneliness and hopelessness in hemodialysis patients. Therapeutic touch treatment method wil lprovide nurses the holistic caregiver role for the feelings of loneliness and hopelessness experienced by the patients. When the literature is scanned, this study is unique because it has not been done before on hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Having hemodialysis treatment for at least 3 months,
* Cognitive patients,
* Having a score of UCLA> 20 and BECK≥4 scoring,
* Involved in the work with us.

Exclusion Criteria:

• Patients using traditional treatment for the disease were not included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
The effect of therapeutic touch on loneliness in hemodialysis patients | Scales are filled after 3 days of application.
  Developed by Russell et al. in 1980, the UCLA Loneliness Scale consists of 20 items, 10 of which are straight and 10 of which are reversed. Each item is scored between 1-4. While calculating the loneliness score, the calculation is made by taking the reverse of the scores given to the items used adversely. The highest score that can be obtained from the scale is 80, and the lowest score is 20. Higher scores indicate that individuals experience more loneliness.
The effect of therapeutic touch on hopelessness in hemodialysis patients | Scales are filled after 3 days of application.
  The scale developed by Beck et al. in 1974 to measure hopelessness consists of 20 items and is scored between 0 and 1. The items in the scale are Emotions and Expectations about the Future (1, 3, 7, 11 and 18), Loss of Motivation (2, 4, 9, 12, 14, 16, 17 and 20), and Hope (5, 6, 8, 10, 13). , 15 and 19) have three sub-dimensions. The lowest score that can be obtained from the scale is 0, the highest score is 20, and a high score indicates a high level of hopelessness.

CONTACTS AND LOCATIONS:
Overall Officials: Songül Karadağ, Principal Investigator — Cukurova University
Locations (2):
- Turkey (Türkiye) (2):
  - ZEHRA, Bayram
  - Zehra Bayram, Osmaniye

IPD SHARING:
Plan to Share IPD: Yes
Results of intervention and control group scales before and after administration (statistical analysis) Introductory characteristics of the participants and participant consent form
Supporting Information: SAP, ICF
Time Frame: Data is continuously available after publication
Access Criteria: Data can be shared publicly
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/